CLINICAL TRIAL: NCT02673398
Title: Phase II Study of Neratinib in Patients 60 and Older With HER2 Positive Metastatic Breast Cancer
Brief Title: Neratinib in Treating Older Patients With Stage IV HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15342; NCI-2015-02282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15342 (Other: City of Hope Medical Center); K12CA001727 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2016-01-21; First posted 2016-02-03 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: HER2 Positive Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — Geriatric Assessment; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (neratinib) (Experimental): Patients receive neratinib 240mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Laboratory Biomarker Analysis; Drug: Neratinib; Other: Pharmacological Study

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Neratinib — Given PO
  Other Names: (2E)-N-(4-((3-chloro-4-((pyridin-2-yl)methoxy)phenyl)amino)-3-cyano-7-ethoxyquinolin-6-yl)-4-(dimethylamino)but-2-enamide; HKI 272; HKI-272; PB 272; PB-272
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies the side effects of and how well neratinib works in treating older patients with stage IV HER2-positive breast cancer. Neratinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety and tolerability of neratinib in adults age 60 or older with locally advanced or metastatic HER2 over-expressing breast cancer.

SECONDARY OBJECTIVES:

I. To describe the full toxicity profile including all grade toxicities measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0.

II. To estimate the rate of all grades of gastrointestinal (GI) toxicities such as diarrhea, nausea, and vomiting.

III. To estimate the rate of dose reduction, delays and discontinuation related to study drug.

IV. To describe pharmacokinetic parameters of neratinib in adults 60 and older. V. To estimate overall response rate (ORR) and clinical benefit rate (CBR) defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

VI. To estimate event free survival (EFS), progression-free survival (PFS) and overall survival (OS).

VII. To evaluate the role of cancer-specific geriatric assessment tool in predicting treatment toxicities.

VIII. To estimate adherence rate to neratinib in older adults (percentage of doses of neratinib taken).

IX. To explore the association of pharmacokinetic (PK) parameters and geriatric assessment findings.

X. To explore if serum biomarkers of aging (interleukin [IL]-6, C-reactive protein [CRP], and D-dimer) are associated with treatment toxicities.

OUTLINE:

Patients receive neratinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* Life expectancy of greater than 12 weeks
* Histologically or cytologically proven metastatic breast cancer (metastases can be proven with imaging results in certain circumstances provided that the initial tumor was demonstrated histologically)
* Stage IV HER2/Neu positive breast cancer patients who failed previous anti-HER2 targeted therapies
* HER2 positivity as defined by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* If HER2 negative by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH), but activating somatic mutations of HER2 gene identified through genomic sequencing including but not limited to the following (Clinical Laboratory Improvement Act [CLIA] certified lab test): missense substitutions (G309A, G309E, S310F, S310Y, S653C, V659E, R678Q, V697L, T733I, L755S, L755P, E757A, D769H, D769Y, D769N, G776V, G776C, V777L, L841V, V842I, R849W, L869R, R896C); insertions/deletions (A775_G776insYVMA aka Y772_A755dup, G776VinsC, G776AinsVGC, G776 insertions, G778_S779insCPG, P780_781insGSP aka G778_P780dup, L755_T759del) and/or HER3 activating mutations; there is no limitation on the number of prior lines of systemic therapy or HER2-targeted therapies (prior neratinib not allowed)
* Both measurable as well as non-measurable disease will be allowed
* Hemoglobin >= 9 g/dL (after transfusion, if necessary) within 4 weeks of pre-registration
* Total bilirubin within normal institutional limits within 4 weeks of pre-registration
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal within 4 weeks of pre-registration
* Creatinine clearance >= 30 mL/min as calculated by Cockcroft-Gault formula within 4 weeks of pre-registration
* Baseline left ventricular ejection fraction LVEF >= 50% as evaluated by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* All grade >= 2 toxicities other than alopecia from prior therapy have resolved by the time of study commencement
* Patient must have completed radiation therapy with adequate recovery of bone marrow and organ functions, before starting neratinib
* Patient with stable or treated brain metastases are eligible; asymptomatic patients with metastatic brain disease who have been on a stable dose of corticosteroids for treatment of brain metastases for at least 14 days are eligible to participate in the study
* Provide written, informed consent to participate in the study and follow the study procedures

Exclusion Criteria:

* Prior treatment with neratinib
* Concurrent usage of other investigational agents, chemotherapy, or hormone therapy; prior chemotherapy, hormonal therapy, targeted therapy, and investigational agents are allowed but all toxicities grade >= 2 must have resolved by the time of study commencement (except alopecia)
* Any major surgery =< 28 days prior to the initiation of investigational products
* Received chemotherapy or biologic therapy =< 3 weeks prior to the start of neratinib
* Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of >= 2, including individuals who currently use digitalis specifically for congestive heart failure), unstable angina, myocardial infarction within 12 month of enrollment or ventricular arrhythmia
* Concurrent use of digoxin due to cardiac disease; corrected QT (QTc) interval >= 450 milliseconds in men and >= 470 milliseconds in women within 2 weeks of registration or known history of QTc prolongation or Torsades de Pointes
* Inability to take oral medication
* Other malignancy within the past 3 years with the exception of: a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) cervix or vulva carcinoma in situ; c) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder, or benign tumors of the adrenal or pancreas
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn?s disease, malabsorption, or grade >= 2 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v.4.0 diarrhea of any etiology at baseline)
* Known clinically active infection with hepatitis B or hepatitis C virus
* Evidence of significant medical illness, abnormal laboratory finding or psychiatric illness/social situations that would, in the investigator?s judgment, makes the patient inappropriate for this study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, Principal Investigator — City of Hope Medical Center
Locations (7):
- United States (7):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

REFERENCES:
- [Derived] Wong CW, Yost SE, Lee JS, Gillece JD, Folkerts M, Reining L, Highlander SK, Eftekhari Z, Mortimer J, Yuan Y. Analysis of Gut Microbiome Using Explainable Machine Learning Predicts Risk of Diarrhea Associated With Tyrosine Kinase Inhibitor Neratinib: A Pilot Study. Front Oncol. 2021 Mar 10;11:604584. doi: 10.3389/fonc.2021.604584. eCollection 2021. PMID 33796451
- [Derived] Yuan Y, Lee JS, Yost SE, Stiller T, Blanchard MS, Padam S, Katheria V, Kim H, Sun C, Tang A, Martinez N, Patel ND, Sedrak MS, Waisman J, Li D, Sanani S, Presant CA, Mortimer J. Phase II study of neratinib in older adults with HER2 amplified or HER2/3 mutated metastatic breast cancer. J Geriatr Oncol. 2021 Jun;12(5):752-758. doi: 10.1016/j.jgo.2021.02.020. Epub 2021 Mar 2. PMID 33663941

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Neratinib): Patients receive neratinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Comprehensive Geriatric Assessment: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
  Neratinib: Given PO
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Neratinib)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 66 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
ECOG performance status [Count of Participants; unit: Participants]
  0 = Fully active, able to carry on all pre-disease performance without restriction | 8
  1 = Restricted in physically strenuous activity but ambulatory and able to do work of a light nature | 17
Hormone receptor status [Count of Participants; unit: Participants]
  Positive | 19
  Negative | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Grade 2 or Higher Toxicities
Description: Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Tables will be created to summarize the toxicities and side effects by organ system, attribution and severity for all participants that receive at least one dose of neratinib. Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for grade 2 or higher toxicities attributed to neratinib.
Time Frame: On treatment, 28 days per cycle up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
percentage of participants | 80 [59 to 93]

2. Secondary Outcome: Count of Participants With Grade 3 or Higher Gastrointestinal (GI) Toxicities Such as Diarrhea, Nausea and Vomiting
Description: Will be graded according to the NCI CTCAE version 4.0. Tables will be created to summarize the toxicities and side effects by organ system, attribution and severity for all participants that receive at least one dose of neratinib.
Time Frame: On treatment, 28 days per cycle up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
Participants
  Diarrhea | 5
  Vomiting | 2
  Abdominal pain | 2
  Nausea | 1

3. Secondary Outcome: Rate of Participants With a Dose Reduction
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for dose reduction.
Time Frame: On treatment, up to 48 months
Population: 9 of 25 patients 36% had a dose reduction.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
percentage of participants | 36 [18 to 57]

4. Secondary Outcome: Rate of Participants Requiring Hospitalizations
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for hospitalizations.
Time Frame: On treatment, up to 48 months
Population: 4 of 25 patients (16%) were hospitalized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
percentage of participants | 16 [5 to 36]

5. Secondary Outcome: Tumor Response Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Complete Response (CR): Disappearance of all target lesions. Lymph node CR is when the lymph node has decreased to less than 10mm in the short axis.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started (including the baseline scan if that is the smallest), and at least a 5mm increase or the appearance of new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Participants are evaluated every 12 weeks, up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
Participants
  Partial Remission | 1
  Stable Disease | 11
  Progressive Disease | 12
  Not assessed | 1

6. Secondary Outcome: Median Progression-free Survival (PFS) in Months
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for PFS. PFS will be estimated using the product limit method of Kaplan and Meier.
Time Frame: From the date treatment begins until the first date on which recurrence, progression or death due to any cause, assessed up to 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
months | 2.6 [2.56 to 5.26]

7. Secondary Outcome: Median Overall Survival (OS)
Description: OS will be estimated using the product limit method of Kaplan and Meier.
Time Frame: Time from start of treatment to death due to any cause, assessed up to 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 25
months | 17.4 [10.3 to NA] — insufficient number of participants with events

8. Secondary Outcome: Cancer-specific Geriatric Assessment Score
Description: The cancer specific geriatric assessment score includes an evaluation of functional status, co-morbidity, cognition, psychological stats, social functioning and support, and nutritional status. It assesses a patient's age, gender, height, weight, cancer type, dosage, number of chemotherapy agents, hemoglobin, hearing, number of falls in past 6 months, able to take own medicine, whether walking is limited, have physical or emotional problems interfered with social activities and serum creatinine.
  Scores can range from 0 to to 1, with a higher score indicating higher risk of chemotherapy toxicity.
  Generalized linear models and graphical methods will be used to explore factors as identified by a cancer-specific geriatric assessment.
Time Frame: At day 0 of treatment
Population: 3 participants did not have complete geriatric assessment data.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 22
scores on a scale | 0.34 [0.19 to 0.59]
Statistical Analysis 1: Comparison: Treatment (Neratinib); Student's t-test was used to assess if geriatric risk score differed depending on whether or not a participant had a dose reduction (mean difference log2 risk = no dose modification - dose modification); Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.82 to 0.01] — Patients with higher risk scores were more likely to require a dose reduction. The lack of significance is most likely due to the small sample size
Statistical Analysis 2: Comparison: Treatment (Neratinib); Linear regression was used to assess whether log2 geriatric toxicity risk score was a risk factor for the number of course completed; Test type: Superiority; p = 0.39, Regression, Linear; Slope = -1.29, Standard Error of Mean 1.44

9. Secondary Outcome: Pharmacokinetics of Steady State Neratinib Concentration Transformed Using a Logarithm Base 2
Description: Least squares regression was used to assess the relationship between steady state neratinib concentration, transformed using a logarithm base 2 transformation, and age
Time Frame: Day 0 to day 15
Population: Only 20 participants had PK data available.
Measure: Mean (Standard Deviation); unit: log2(ng/mL)
Arm/Group | Treatment (Neratinib)
Number analyzed (Participants) | 20
log2(ng/mL) | 4.7 (1.09)
Statistical Analysis 1: Comparison: Treatment (Neratinib); Least squares regression was used to assess the relationship between steady state neratinib concentration and age; Test type: Superiority; p = 0.03, Regression, Linear; Slope = -0.093, Standard Error of Mean 0.0398 — The older the participant the lower the steady state value
Statistical Analysis 2: Comparison: Treatment (Neratinib); Least squares regression was used to determine if geriatric toxicity risk score at baseline was predictive of steady state neratinib concentration; Test type: Superiority; p = 0.57, Regression, Linear; Slope = 1.4, Standard Deviation 2.39 — Geriatric risk score was not predictive of steady state concentration

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 18 months
Description: All serious adverse events are reported regardless of attribution and grade. Count of participants experiencing grade 2, 3, 4, or 5 other adverse events possibly, probably, or definitely attributed to neratinib are reported (after removing serious adverse events from the toxicity dataset).
Arm/Group | Treatment (Neratinib)
All-Cause Mortality (participants affected / at risk) | 16/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neratinib) (N=25)
Pericardial tampo (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Weight loss (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
T7 mets with spinal cord compression (Musculoskeletal and connective tissue disorders) | 1
Death (General disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neratinib) (N=25)
Anemia (Blood and lymphatic system disorders) | 4
Lymphocyte count decreased (Blood and lymphatic system disorders) | 6
White blood cell count decreased (Blood and lymphatic system disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Anorexia (General disorders) | 3
Dehydration (General disorders) | 2
Fatigue (General disorders) | 3
Generalized muscle weakness (General disorders) | 1
Weight loss (General disorders) | 1
Acute kidney injury (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin laceration (Skin and subcutaneous tissue disorders) | 1
Ejection fraction decreased (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Hypoalbuminemia (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02673398/Prot_SAP_000.pdf